CLINICAL TRIAL: NCT04828031
Title: Vitamin D Regulation of α4β7+ B Cell Immunophenotypes and Mucosal Antibody Response to Commensal Gut Bacteria in Patients With Inflammatory Bowel Disease
Brief Title: Vitamin D Regulation of Gut Specific B Cells and Antibodies Targeting Gut Bacteria in Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Principal Investigator, John Gubatan, Fellow in Gastroenterology, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-60958
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Inflammatory Bowel Diseases; Ulcerative Colitis; Crohn Disease
Keywords: Gut Microbiome, Vitamin D, Dysbiosis, Inflammation
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease; Dysbiosis; Inflammation | interventions — Vitamin D

STUDY DESIGN:
Intervention Model Description: Open label prospective clinical trial with vitamin D 50,000 IU PO every week for 12 weeks in patients with inflammatory bowel disease (IBD) with 25(OH)D ≤ 25 ng/mL
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vitamin D 50,000 IU PO every week (Experimental): Vitamin D 50,000 IU PO every week for 12 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Patient with inflammatory bowel disease who have low vitamin D (25(OH)D less than or equal to 25 ng/mL) will take Vitamin D 50,000 IU by mouth every week for 12 weeks. Patients will fill out questionnaires to document disease activity score (HBI or Mayo score and sIBDQ) and have blood and stool samples collected before (Week 0), during (Week 8) and after (Week 12) vitamin D intervention.

SUMMARY:
Specific Aim 1: Characterize the effects of vitamin D treatment on expression of α4β7 on B cells in patients with inflammatory bowel disease (IBD).

Specific Aim 2: Determine the effects of vitamin D treatment on fecal immunoglobulins, percentage of Ig-coated gut bacteria, gut microbiome composition (global and bound by immunoglobulins) in patients with IBD and the association of these parameters with change in α4β7+ B cells .

Specific Aim 3: Compare BCR repertoire (BCR clonotypes, immunoglobulin heavy chain gene (IGHV), and isotype usage) between α4β7+ and α4β7- B cells in patients with IBD and identify α4β7+ BCR clonotypes associated with Ig-bound gut bacteria .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years or older) with inflammatory bowel disease (ulcerative colitis or Crohn's disease)
* Low serum vitamin D (25(OH)D ≤ 25 ng/mL
* Not currently on high dose vitamin D supplementation
* No prior bowel resections
* No antibiotic use in past 3 months.

Exclusion Criteria:

* Patients less than 18 years old
* No diagnosis of IBD
* Serum 25(OH)D > 25 ng/mL
* Patients already on vitamin D supplementation
* Prior history of bowel surgery (colectomy or small bowel resections)
* Recent antibiotic use in past 3 months
* Renal Dysfunction
* History of Hypercalcemia
* History of HIV
* History of IgA deficiency
* History of Common Variable Immunodeficiency (CVID)
* Active C. diff infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Reduction in α4β7+ B cells by 20% | Week 12
  Expression of gut tropic integrin α4β7+ on B cells assessed at gene expression level (single cell transcriptomics) and protein level (cytometry)
Reduction in immunoglobulin coating of commensal gut bacteria by 20%. | Week 12
  Immunoglobulin coating of gut bacteria will be measured from stool samples using Ig-Seq

SECONDARY OUTCOMES:
Increase in serum vitamin D (25(OH)D levels by 10 ng/mL | Week 12
  25(OH)D will be measured from serum by standard laboratory assay (HPLC)
Decrease in disease activity index scores by 50% | Week 12
  Disease activity index scores will be measured by Harvey Bradshaw Index in Crohn's disease patients and Mayo Score disease activity index in ulcerative colitis patients
Decrease cohort mean fecal calprotectin or C-reactive protein (CRP) by 50%. | Week 12
  Fecal calprotectin will be measured from stool samples. CRP will be measured from plasma

CONTACTS AND LOCATIONS:
Overall Officials: John Mark Gubatan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] de Souza HSP, Fiocchi C, Iliopoulos D. The IBD interactome: an integrated view of aetiology, pathogenesis and therapy. Nat Rev Gastroenterol Hepatol. 2017 Dec;14(12):739-749. doi: 10.1038/nrgastro.2017.110. Epub 2017 Aug 23. PMID 28831186
- [Background] Caruso R, Lo BC, Nunez G. Host-microbiota interactions in inflammatory bowel disease. Nat Rev Immunol. 2020 Jul;20(7):411-426. doi: 10.1038/s41577-019-0268-7. Epub 2020 Jan 31. PMID 32005980
- [Background] Rengarajan S, Vivio EE, Parkes M, Peterson DA, Roberson EDO, Newberry RD, Ciorba MA, Hsieh CS. Dynamic immunoglobulin responses to gut bacteria during inflammatory bowel disease. Gut Microbes. 2020 May 3;11(3):405-420. doi: 10.1080/19490976.2019.1626683. Epub 2019 Jun 16. PMID 31203722
- [Background] Castro-Dopico T, Dennison TW, Ferdinand JR, Mathews RJ, Fleming A, Clift D, Stewart BJ, Jing C, Strongili K, Labzin LI, Monk EJM, Saeb-Parsy K, Bryant CE, Clare S, Parkes M, Clatworthy MR. Anti-commensal IgG Drives Intestinal Inflammation and Type 17 Immunity in Ulcerative Colitis. Immunity. 2019 Apr 16;50(4):1099-1114.e10. doi: 10.1016/j.immuni.2019.02.006. Epub 2019 Mar 12. PMID 30876876
- [Background] Gubatan J, Chou ND, Nielsen OH, Moss AC. Systematic review with meta-analysis: association of vitamin D status with clinical outcomes in adult patients with inflammatory bowel disease. Aliment Pharmacol Ther. 2019 Dec;50(11-12):1146-1158. doi: 10.1111/apt.15506. Epub 2019 Oct 24. PMID 31647134
- [Background] Gubatan J, Mitsuhashi S, Zenlea T, Rosenberg L, Robson S, Moss AC. Low Serum Vitamin D During Remission Increases Risk of Clinical Relapse in Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2017 Feb;15(2):240-246.e1. doi: 10.1016/j.cgh.2016.05.035. Epub 2016 Jun 4. PMID 27266980
- [Background] Gubatan J, Moss AC. Vitamin D in inflammatory bowel disease: more than just a supplement. Curr Opin Gastroenterol. 2018 Jul;34(4):217-225. doi: 10.1097/MOG.0000000000000449. PMID 29762159
- [Background] Sigmundsdottir H, Pan J, Debes GF, Alt C, Habtezion A, Soler D, Butcher EC. DCs metabolize sunlight-induced vitamin D3 to 'program' T cell attraction to the epidermal chemokine CCL27. Nat Immunol. 2007 Mar;8(3):285-93. doi: 10.1038/ni1433. Epub 2007 Jan 28. PMID 17259988
- [Background] Gubatan J, Rubin SJS, Bai L, Haileselassie Y, Levitte S, Balabanis T, Patel A, Sharma A, Sinha SR, Habtezion A. Vitamin D Is Associated with alpha4beta7+ Immunophenotypes and Predicts Vedolizumab Therapy Failure in Patients with Inflammatory Bowel Disease. J Crohns Colitis. 2021 Dec 18;15(12):1980-1990. doi: 10.1093/ecco-jcc/jjab114. PMID 34180967